CLINICAL TRIAL: NCT02355626
Title: Prognosis of Anxiety in Intensive Care Unit
Acronym: PAN-ICU
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Tarek Sharshar, Tarek SHARSHAR, MD, PHD, Assistance Publique - Hôpitaux de Paris
Other Study IDs: 12-PANICU
Record Dates: First submitted 2014-11-14; First posted 2015-02-04 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Anxiety
Keywords: Anxiety; level of anxiety; delirium; agitation; tools for measuring anxiety; neuroendocrine system
MeSH Terms: conditions — Anxiety Disorders; Delirium; Psychomotor Agitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Anxiety is commonly considered as an epiphenomenon of the cognitive and emotional response to a threat. Anxiety is a consequence of the reciprocal interaction between stress and the neuroendocrine, autonomic and immune systems. A systematic and circumstantial assessment of anxiety in critically ill patients has never been done. Our hypothesis is that high levels of anxiety at ICU admission are associated with death or the occurrence of one or more organ failure during the first 7 days, and that anxiety should be considered as a "warning sign" in critically ill patients.

DETAILED DESCRIPTION:
Multicentre prospective study. Demographic data, diagnosis, severity scores and vital signs will be assessed at admission.

Within the first 12 hours, and at day 4 and day 7, anxiety will be assessed by the STAI scale, Geriatric Anxiety Inventory (GAI) scale, and a specific questionnaire assessing anxiety in the intensive care (REAX). Visual Analogue Scale (VAS) scoring for anxiety, starvation, thirst, pain and dyspnoea will be collected daily. Anxiety and depression will be evaluated by the Hospital Anxiety and Depression Scale (HADS) on day 7. Patients will be assessed by psychologists or trained doctors, the team in charge of the patient will not be aware of the result of this evaluation.

Clinical and biological data regarding the hemodynamic, neurological, respiratory and renal status will be collected from admission to day 7, as well as parameters required for computing the Sequential Organ Failure Assessment (SOFA) score.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the ICU
* Patient without delirium at admission (assessed using the CAM-ICU score)

Exclusion Criteria:

* Severe hearing impairment or poor understanding of French language
* History of serious psychiatric illness
* Comatose or sedated patient at admission
* Diagnosis of voluntary self-poisoning, or polytrauma at admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients, not comatose and not confused
Sampling Method: Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of death or organ failure. | 7 days

SECONDARY OUTCOMES:
1-Occurrence of shock, delirium, or stress-related complications (upper gastrointestinal bleeding, acute coronary syndrome) | 7 days
Severity of an ongoing organ failure (maximum SOFA score) | 7 days
Assessment of anxiety according to State Trait Anxiety Inventory score (STAI) | 7 days
Assessment of anxiety according to REAX score | 7 days
Assessment of anxiety according to the Visual Analog Scale (VAS) | 7 days
Assessment of Geriatric Anxiety Inventory score (GAI) | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Sharshar, MD, PHD, Principal Investigator — General intensive care unit Raymond Poincaré Hospital, 92380 Garches, France
Locations (1):
- General intensive care unit Raymond Poincaré Hospital, Garches, Hauts-de-seine, France

REFERENCES:
- [Derived] Mazeraud A, Turc G, Sivanandamoorthy S, Porcher R, Stoclin A, Antona M, Polito A, Righy C, Bozza FAB, Siami S, Sharshar T. Association of Lack of Fear of Dying With New Organ Failure: Results of a Multicenter Prospective Cohort Study. Am J Crit Care. 2024 Jan 1;33(1):36-44. doi: 10.4037/ajcc2024517. PMID 38161174
- [Derived] Mazeraud A, Polito A, Sivanandamoorthy S, Porcher R, Heming N, Stoclin A, Hissem T, Antona M, Blot F, Gaillard R, Chretien F, Annane D, Bozza FAB, Siami S, Sharshar T; Groupe d'Explorations Neurologiques en Reanimation (GENER). Association Between Anxiety and New Organ Failure, Independently of Critical Illness Severity and Respiratory Status: A Prospective Multicentric Cohort Study. Crit Care Med. 2020 Oct;48(10):1471-1479. doi: 10.1097/CCM.0000000000004495. PMID 32931190